CLINICAL TRIAL: NCT05910554
Title: Investigation of the Efficacy of Metformin Therapy on Pulmonary Sarcoidosis Phase II Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Investigation of the Efficacy of Metformin Therapy on Pulmonary Sarcoidosis
Acronym: MetforminTOP
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Many of sarcoidosis patients in this area already taking metformin
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00105681
Record Dates: First submitted 2023-06-06; First posted 2023-06-18 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Sarcoidosis, Pulmonary
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Metformin; Glyburide; Cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Metformin capsules will be encapsulated by the Investigational Drug Services to blind study participants and providers, as well study personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Patients randomized to metformin will be assigned the active arm.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Patients randomized to cellulose will be assigned the placebo arm.
  Interventions: Drug: Cellulose

INTERVENTIONS:
Drug: Metformin — Patients randomized to metformin will be assigned the active arm.
  Other Names: glyburide
  Arms: Active
Drug: Cellulose — Patients randomized to cellulose will be assigned the placebo arm.
  Other Names: cellulose powder
  Arms: Placebo

SUMMARY:
This is a double blinded, randomized, placebo controlled clinical trial of 40 participants with pulmonary sarcoidosis.

Primary Objective: To assess the steroid-sparing efficacy and safety of oral metformin therapy in participants with confirmed progressive pulmonary sarcoidosis for participants with steroid dependent disease.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy of Metformin therapy in terms of steroid-sparing efficacy for sarcoidosis patients with steroid-dependent disease. Given that the morbidity and mortality has proven to be significant in patients with sarcoidosis, we believe there is unprecedented opportunity for improved clinical outcomes if the right interventional agent can be identified. In choosing steroid-sparing effect as the primary outcome, we will be able to detect changes in clinical outcomes that are important to patients and to the scientific community. We anticipate that these improvements will reduce or resolve the necessity of immunosuppressant therapy in these participants.

At least 40 participants will be randomized in equal proportion to metformin or placebo. Twenty completed participants per arm provide 80% power to reject (one-sided type I error of 5%) the null hypothesis that mean daily steroid use in the placebo treated group is less than in the metformin treated group using analysis of covariance adjusting for baseline average steroid use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with sarcoidosis as defined by the ATS/ERS/WASOG statement on sarcoidosis as defined by the clinical presentation consistent with sarcoidosis, as well as biopsy demonstrating granulomas, and no alternative for the cause of the granulomas, such as tuberculosis for at least one year prior to randomization. Tuberculosis must be ruled out by negative histology and culture.
2. Patients must be symptomatic of pulmonary sarcoidosis with FVC 45-85%
3. Steroid dosage of >10mg of prednisone for at least 6 months

Exclusion Criteria:

1. Inability to obtain consent
2. Age less than 18 years of age
3. Female participants of childbearing potential not willing use one of the following methods of birth control for the duration of the study and 90 days after study completion: condoms, sponge, foams, jellies, diaphragm, or non-hormonal intrauterine device, a vasectomized sole partner or abstinence. Females of childbearing potential must have a negative urine pregnancy test at screening visit
4. FVC predicted value is < 45%.
5. Creatine clearance of <30%.
6. History of idiopathic Lactate ≥ 2.2 mmol/L or acidosis on study baseline metabolic profile
7. End-stage fibrotic pulmonary disease
8. Significant underlying liver disease
9. Allergy or intolerance to metformin
10. Allergy or intolerance to albuterol
11. Poor venous access for obtaining blood samples
12. Significant disorder, other than sarcoidosis, that would complicate the treatment evaluation, such as respiratory, cardiac, renal, neurologic, musculoskeletal or seizure disorders.
13. Use of an investigational drug within 30 days prior to screening or within 5 half-lives of the agent, whichever is longer.
14. Currently receiving >40mg prednisone.
15. ALT or AST ≥5 times upper limit of normal (ULN).
16. Leukopenia, as defined by WBC <3.0 cells/mm3 or absolute neutrophil count <1000 mm3
17. Breast feeding.
18. If patient is on immunomodulators, they must be on regimen for ≥3-month period and on a stable dose for ≥ 4 weeks.
19. Most recent nuclear medicine scan or echocardiogram (if done), demonstrating cardiac ejection fraction <35%
20. Participant has persistent or active infections requiring hospitalization or treatment with antibiotics, antiretrovirals, or antifungals within 30 days of baseline. Minocycline and doxycycline are not considered antibiotics when used to treat sarcoidosis.
21. Any significant finding in the patient's medical history or physical or psychiatric exam prior to or after randomization that, in the opinion of the investigator, would affect patient safety or compliance or ability to deliver the study drug according to protocol.
22. On medications that, in the opinion of the investigator, would affect patient safety when taken with metformin
23. History of or receiving treatment for pulmonary hypertension. Receiving biologic medication within the 6 months prior to screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the steroid-sparing efficacy and safety of oral metformin therapy in patients with progressive pulmonary sarcoidosis. | 24 weeks
  Mean daily oral corticosteroid dose post protocol-driven steroid taper at 24-weeks after randomization.

SECONDARY OUTCOMES:
To compare cumulative total steroid use between those randomized to metformin or placebo | 24 weeks
  • Average dose and cumulative total steroid use in the 24-week study horizon.

IPD SHARING:
Plan to Share IPD: No
No HIPAA data will be provided.